CLINICAL TRIAL: NCT06512714
Title: Estimating the Burden of Mycetoma: A Retrospective Analysis of Hospital Records
Brief Title: Mycetoma Retrospective Data Collection
Status: Recruiting | Type: Observational
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Cheikh Anta Diop University, Senegal (Other); Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Sponsor
Other Study IDs: DNDi-OBS-03-MYC
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Mycetoma
MeSH Terms: conditions — Mycetoma | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: A diagnosis of mycetoma in a medical, radiologic, or laboratory record. — For each patient, data will be extracted for each clinical, laboratory or radiologic visit related to the condition that may meet this study's case definition.

SUMMARY:
The goal of this retrospective observational study is to describe mycetoma cases detected in health care facilities in India and Senegal in a 10-year period. The main objectives are to:

* Determine the number of mycetoma cases diagnosed per year and trends over time.
* Describe characteristics of diagnosed mycetoma cases.

  1. Describe demographic characteristics of patients with mycetoma.
  2. Describe clinical characteristics of patients with mycetoma upon initial presentation and over time.
* Assess etiology of mycetoma cases.
* Characterize clinical management of mycetoma cases.

  1. Characterize approaches to diagnosis of mycetoma.
  2. Investigate types and durations of treatments (including medical and surgical approaches) utilized to treat mycetoma cases.
  3. Describe clinical outcomes among patients with mycetoma.

The study team will review all available medical, laboratory and radiologic records of identified mycetoma cases and use data collection forms to extract relevant data.

DETAILED DESCRIPTION:
Mycetoma is a poorly understood neglected tropical disease which disproportionately affects the poorest of the poor and is associated with substantial morbidity. The disease presents a multitude of diagnostic and management challenges; in particular, effective treatments for eumycetoma, the fungal and least understood form of the disease are lacking. DNDi and partners aim to conduct late-phase clinical trials on a promising new pharmacologic treatment for eumycetoma, but substantial knowledge gaps preclude such trials. These knowledge gaps include data on the burden, distribution, causative agents, clinical presentation, natural history, and common approaches to diagnosis and treatment of mycetoma in endemic countries.

This study, a retrospective review of mycetoma cases, aims to generate such data from several countries suggested by preliminary data to potentially be good candidate clinical trial sites.

ELIGIBILITY:
Inclusion Criteria:

* Any patient given a diagnosis of mycetoma in a medical, radiologic, or laboratory record.

Exclusion Criteria:

* Patients with illegible or inaccessible health records.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient given a diagnosis of mycetoma in a medical, radiologic, or laboratory record.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Presence of mycetoma disease as evidenced by patient diagnosis | Over 10 years
  Sources: Medical records and/or laboratory records and/or radiologic records.

SECONDARY OUTCOMES:
Lesion size in centimeters | Over 10 years
  Sources: Medical records and laboratory records
Presence of mycetoma disease after treatment or surgery | Over 10 years
  Sources: Medical records and laboratory records

CONTACTS AND LOCATIONS:
Overall Officials: Doudou Sow, PhD, Principal Investigator — Université Gaston Berger; Shivaprakash M Rudramurthy, M.D, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (2):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India
- Universite Cheikh Anta Diop de Dakar, Dakar, Senegal

IPD SHARING:
Plan to Share IPD: Yes
Through Drugs for Neglected Diseases Initiative (DNDi) and open data sharing platforms. The data may be obtained by sending a request to DNDi, de-identified or aggregated data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Within 24 months of last subject last visit
Access Criteria: Data Requestors seeking individual participant level data will enter into an appropriate agreement or terms of use.
URL: http://dndi.org